CLINICAL TRIAL: NCT03520244
Title: Understanding the Relationship Between the MicrobiOme, Vitality and Exercise in Celiac Disease (MOVE-C)
Brief Title: A 12-week Exercise Program for Adults With Celiac Disease
Acronym: MOVE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB16-1774
Record Dates: First submitted 2017-02-21; First posted 2018-05-09 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-04

CONDITIONS: Celiac Disease
Keywords: Microbiome; High intensity interval training; Exercise; Holistic education; Quality of life; Fatigue
MeSH Terms: conditions — Celiac Disease; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups in parallel for the duration of the study. One group is interventional (exercise + education sessions). This group will be evaluated in parallel against a wait-list control group.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are masked to participant group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + Holistic Education (Experimental): A 12-week exercise program with 6 bi-weekly education sessions.
  Interventions: Behavioral: Exercise + Holistic Education
- Wait list control (No Intervention): Participants in the control group will be offered the exercise + education sessions after the study is complete.

INTERVENTIONS:
Behavioral: Exercise + Holistic Education — The exercise group will undertake a 12-week supervised progressive high intensity interval training program supplemented with 6 bi-weekly group-based holistic education sessions.
  Arms: Exercise + Holistic Education

SUMMARY:
Engagement in regular physical activity (PA) is associated with a range of physical and psychological benefits among chronic disease populations. Celiac disease is a chronic autoimmune condition that requires strict adherence to a gluten-free diet (GFD) for the best medical outcomes, as well as to prevent detrimental health outcomes including bloating, diarrhea, constipation, and increased risk of intestinal cancers and osteoporosis. Despite following a GFD, individuals with celiac disease often report dissatisfaction with the diet, are less likely to engage in social activities, can have an imbalance in gut bacteria and up to 30% still report negative symptoms (e.g., gastro-intestinal upset). Furthermore, preliminary research revealed that rates of PA among those with celiac disease are dismal, with the majority of participants failing to engage in regular PA. The purpose of this pilot research project is to examine the effects of a 12-week structured exercise program on inactive adults with celiac disease. It is anticipated that compared to those in a wait-list control condition, participants who engage in the 12-week exercise program will report greater improvements in quality of life and experience improved balance of gut bacteria. The findings from this project may reveal an additional strategy to optimize health while living with celiac disease. In addition, results from this study will provide essential pilot data that will inform a grant application for a larger clinical trial to further investigate the role of exercise in the promotion of health and well-being among those with celiac disease.

DETAILED DESCRIPTION:
Background & Rationale:

Engagement in regular physical activity (PA) is associated with a range of physical and psychological benefits among chronic disease populations. Quality of life (QoL) is significantly higher among people with cancer, depression and coronary heart disease who engage in PA on a regular basis. Risk of other chronic diseases such as type 2 diabetes is significantly reduced when people engage in regular PA. In addition, findings from a recent intervention study revealed that after engaging in a 12-week structured exercise program, cancer survivors had improvements in physical functioning, and reductions in fatigue and tiredness.

One chronic disease population that could particularly benefit from engaging in regular PA is people with celiac disease. Celiac disease is a chronic autoimmune condition and the incidence has increased 4 to 5 times over the past 50 years. Strict adherence to a gluten-free diet (GFD) is currently the only treatment for preventing both short- and long-term consequences from celiac disease (e.g., infertility, intestinal cancers, osteoporosis). Unfortunately, preliminary research revealed that rates of PA among those with celiac disease are dismal, with the majority of participants failing to engage in regular PA. Further, following a strict GFD alone may not be sufficient to effectively manage the disease, and can be associated with detrimental outcomes including reduced QoL. Despite following a GFD, individuals with celiac disease report high treatment burden, lower social engagement, fatigue, altered gut microbiota, and up to 30% still report negative symptoms (e.g., gastro-intestinal upset). Given the benefits of engagement in regular PA for other chronic disease populations, helping people with celiac disease become more physically active may lead to improvements in QoL and physiological outcomes.

High-Intensity Interval Training (HIIT) has been found to be appropriate for those with lifestyle-induced chronic diseases, including type 2 diabetes, atherosclerotic cardiovascular disease and metabolic syndrome. HIIT involves repeated bouts of high intensity effort followed by varied recovery times and can be easily modified for people of all fitness levels and chronic conditions. For example, Jung and colleagues reported on the benefits of HIIT for people with pre-diabetes and found that compared to participants engaging in moderate intensity continuous training, participants who engaged in regular bouts of HIIT exercise had better adherence to independent exercise. Martinez et al. found that participants who engaged in shorter interval training (e.g., HIIT), reported more pleasure and enjoyment of the exercise when compared to heavy, continuous or longer interval exercise. In addition to improvements in behavioural outcomes, Denou and colleagues recently found that HIIT also led to improvements in the gut microbiota of mice with diet induced obesity. Given that people with celiac disease are at increased risk of metabolic syndrome and are likely to have gut dysbiosis (imbalance in gut microorganisms), it is anticipated that HIIT may lead to improvements in key psychosocial (e.g., QoL) and behavioural outcomes (i.e., exercise adherence). Further, key markers of metabolic syndrome and balance in the gut microbiota may be positively impacted.

Study aims:

The proposed study is an innovative examination of the effects of exercise on physiological and patient-reported outcomes among people with celiac disease. Specifically, we will explore the effects of a 12-week HIIT and lifestyle intervention on QoL, gut microbiota profile, independent PA, fatigue, and markers of metabolic syndrome (waist circumference, fasting glucose, serum lipids, blood pressure) among people with celiac disease who are currently sedentary (i.e., not meeting Canada's PA Recommendations (150 minutes of weekly activity at a moderate intensity or greater).

Exercise program:

The 12-week exercise program will entail two 60-minute structured group exercise sessions per week. As participants will not be meeting the recommended guidelines for weekly PA, workouts will be progressive in nature and an initial conditioning phase will be integrated into the 12-week program. Participants will begin with 20-30 minute exercise sessions and progress to 40-60 minute sessions over the course of 12 weeks. Each class will consist of warm-up, training period, cool-down and flexibility sections. Participants will have the option of using various pieces of equipment, including stationary bikes, treadmills and ellipticals. All participants will wear heart rate monitors in order to monitor workout intensity. Participants' programs will be designed by a Canadian Society of Exercise Physiology (CSEP) Certified Exercise Physiologist® and exercise classes will be supervised by a CSEP-Certified Personal Trainer®.

Education sessions:

Participants in the exercise condition will participate in 30-minute bi-weekly group education sessions. Education will pertain to learning about the importance of following a nutritious, whole foods-based GFD to effectively manage celiac disease, communication strategies, effective sleep hygiene practices, and strategies to overcome barriers to following a strict GFD. Participants will also be taught behaviour change skills based on the theoretically-based group-mediated cognitive behavioural (GMCB) approach. GMCB interventions teach participants how to self-monitor daily activity, set goals and overcome barriers to regular PA. To prevent dependence on the group, self-regulation becomes a greater emphasis over the course of the GMCB sessions. Previous GMCB interventions have lead to greater improvements in frequency of PA, long-term adherence, fitness, self-efficacy for mobility, and barrier self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years+, diagnosed with celiac disease (blood test and/or biopsy), lives in the Calgary area, inactive (engage in exercise on 2 or less days of the week for 30 mins or less)

Exclusion Criteria:

* medical condition preventing engagement in progressive high intensity interval training, unable to attend exercise sessions at the University 2x/week for 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Celiac Disease Quality of Life (CD-QoL) | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in Celiac Disease Quality of Life (CD-QoL)
Microbiome | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in balance of gut microbiome assessed through stool samples analysis

SECONDARY OUTCOMES:
Adherence to a Gluten-free Diet | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change on the Celiac Dietary Adherence Test
Exercise behaviour | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in independent exercise behaviour through the Godin Leisure Time Exercise Questionnaire
Self-regulatory efficacy - exercise | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in self-regulatory efficacy to exercise
Self-regulatory efficacy - gluten-free diet | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in self-regulatory efficacy to eat a strict gluten-free diet
Sleep quality | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change on the Pittsburg Sleep Quality Index
Gastrointestinal symptoms | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change on the Gastrointestinal Symptom Rating Scale (CeD-GSRS). This scale consists of 10 items that correspond to intensity, frequency, duration and impact on daily living. Outcomes are rated from 1, no discomfort at all, to 7, very severe discomfort, and are combined to compute a mean score.
Self-compassion - Short form | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in self-compassion using the Self-Compassion Scale Short Form (SCS-SF). This scale consists of 12 items with answers ranging from 1 (Almost Never) to 5 (Always). A mean self-compassion score is calculated by taking the reverse score of the negative items prior to calculating the mean.
Waist circumference | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in waist circumference in centimeters
Fasting glucose | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in fasting blood glucose
Serum lipids | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in serum lipids
Blood pressure | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of change in blood pressure following the Canadian Physical Activity Fitness and Lifestyle Appraisal (CPAFLA) protocols.

OTHER OUTCOMES:
Body composition | Baseline, Immediately Post Program and 3 Months After Program
  Assessment of %body fat and % muscle mass through dual-energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: S. Nicole Culos-Reed, PhD, Principal Investigator — University of Calgary; A. Justine Dowd, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowd AJ, Kronlund L, Warbeck C, Parmar C, Daun JT, Wytsma-Fisher K, Reimer RA, Millet G, Fung T, Culos-Reed SN. Effects of a 12-week HIIT + group mediated cognitive behavioural intervention on quality of life among inactive adults with coeliac disease: findings from the pilot MOVE-C study. Psychol Health. 2022 Apr;37(4):440-456. doi: 10.1080/08870446.2021.1921774. Epub 2021 May 26. PMID 34038293
- [Derived] Warbeck C, Dowd AJ, Kronlund L, Parmar C, Daun JT, Wytsma-Fisher K, Millet GY, Schick A, Reimer RA, Fung T, Culos-Reed SN. Feasibility and effects on the gut microbiota of a 12-week high-intensity interval training plus lifestyle education intervention on inactive adults with celiac disease. Appl Physiol Nutr Metab. 2021 Apr;46(4):325-336. doi: 10.1139/apnm-2020-0459. Epub 2020 Sep 22. PMID 32961065